CLINICAL TRIAL: NCT05987319
Title: Feasibility Study to Collect and Assess Safety Data for a Radiofrequency Microneedling Device for Electrocoagulation and Hemostasis of Soft Tissues for Dermatologic Conditions.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYN20-RF-MN-02
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Wrinkle; Fine Lines; Crepey Skin; Acne Scars; Active Acne; Enlarged Pores; Stretch Mark; Loose Skin
MeSH Terms: conditions — Striae Distensae; Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- General Treatment (Experimental): Subjects will receive treatment on the face, neck and/or body for conditions such as but not limited to wrinkles, fine lines, crepey skin, acne scars, active acne, enlarged pores, stretch marks or loose skins.
  Interventions: Device: RadioFrequency Microneedling Device
- Split-face treatment (Experimental): Subjects will receive split-face treatments where each side of the face may be treated with different tips.
  Interventions: Device: RadioFrequency Microneedling Device

INTERVENTIONS:
Device: RadioFrequency Microneedling Device — RadioFrequency device will be used for the treatment of dermatologic conditions.

SUMMARY:
The goal of the Potenza device used in this study is to collect clinical data for dermatologic conditions in which electrocoagulation and hemostasis is a viable mechanism for means of improvement.

DETAILED DESCRIPTION:
Up to 12 subjects will be enrolled at 1 study center. Subjects will be enrolled into 2 groups. Group A will receive treatments on the face, neck, and/or body. Group B will receive split-face treatments where each side of the face may be treated with different tips. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 5 treatments.

ELIGIBILITY:
Inclusion Criteria:

* A healthy, non-smoking male or female between the age of 22-65 years old.
* Fitzpatrick skin type I to VI.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 1 month prior to entering this study.
* The subject has a pacemaker.
* The subject had previous use of gold thread skin rejuvenation.
* The subject has a cut, wound, or infected skin on the area to be treated (but skin eruptions may be treated).
* The subject has a metal implant that interferes with the transmission of energy to the electrical field.
* The subject has any embedded electronic devices that give or receive a signal.
* The subject has Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant.
* The subject is allergic to adhesives such as glues on medical tape: they should be alerted that a rash may occur on the neutral electronic monitoring pad (NEM or neutral pad) site, and an over-the-counter preparation may be used to treat the area.
* The subject is allergic to gold.
* The subject has an unrealistic expectation of the results: this is not plastic surgery, and all subjects should be fully informed of the treatment's expected results.
* The subject has nerve insensitivity to heat in the treatment area or in the neutral pad placement area.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated: this treatment will be ineffective.
* The subject has used Accutane (isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it brittle.
* The subject is taking aspirin or are currently taking antiplatelets, thrombolytics, anti- inflammatories or anticoagulants.
* The subject has a history of bleeding coagulopathies.
* The subject is allergic to topical anesthetic.
* The subject has any of the following conditions:

  * Diabetes
  * Epilepsy
  * Autoimmune disease
  * Herpes simplex
  * HIV
  * Hypertension
  * Dermatitis
* The subject has keloid formation propensity.
* Subjects with electronic implants such as cardiac defibrillator. It may interfere with operation of electronic implants or damage the implants, causing risks.
* The subject has any condition or is in a situation which in the investigator's opinion may put the subject at significant risk, may confound study results or may interfere.

significantly with the subject's participation.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
% of subjects satisfied with treatments. | 30 days post last treatment
  % of subjects satisfied with the treatment will the reported at the 30 days follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Cynosure, Inc., Westford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No